CLINICAL TRIAL: NCT06893796
Title: A Phase Ia Clinical Trial Aimed at Evaluating the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic (PK/PD) Characteristics of Single Dose of Telpegfilgrastim Injection in Healthy Premenopausal Non-pregnant Women
Brief Title: Safety, Tolerability, and PK/PD of Telpegfilgrastim in Premenopausal Non-pregnant Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PG-4-1-002
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia
Keywords: PEG-rhG-CSF; Telpegfilgrastim Injection
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Group 2 (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Group 3 (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection

INTERVENTIONS:
Drug: Telpegfilgrastim Injection — Telpegfilgrastim Injection,0.25mg, s.c.,day 1 single dose .
  Arms: Group 1
Drug: Telpegfilgrastim Injection — Telpegfilgrastim Injection,0.5mg, s.c.,day 1 single dose .
  Arms: Group 2
Drug: Telpegfilgrastim Injection — Telpegfilgrastim Injection,1mg, s.c.,day 1 single dose .
  Arms: Group 3

SUMMARY:
This is an open-label, Phase Ia clinical study to evaluate the safety, tolerability, and pharmacokinetic/pharmacodynamic (PK/PD) characteristics of single dose of telpegfilgrastim injection in healthy premenopausal non-pregnant women. It plans to enroll 18 healthy premenopausal non-pregnant female.,). Participants will be enrolled sequentially according to their screening numbers in the following three dose groups:0.25mg, 0.5mg, and 1mg, with 6 participants in each dose group. Each participant will undergo a screening period (-2 weeks to -2 days), a baseline phase (D-1, the day before the first dose), and a post-dosing observation period (Day 1 to Day 21), and adverse event, vital signs, physical examination, laboratory tests,and PK&PD will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. The participants is able to understand and comply with the contents, requirements, and restrictions of the protocol, complete the study as required by the protocol, and is fully aware of the possible adverse reactions, voluntarily signing the informed consent form before enrolling the trial.
2. Female, aged between 18 and 45 years old (inclusive of 18 and 45 years).
3. Body Mass Index (BMI) ≥ 18.5 and < 28.0 kg/m², weight ≥ 45 kg.
4. At the screening visit and before the first dose on Day 1, a comprehensive physical examination is conducted, including general physical examination, vital signs (pulse between 50 and 100 bpm at rest, systolic blood pressure between 90 and 139 mmHg, diastolic blood pressure between 50 and 89 mmHg, inclusive of the critical values), laboratory tests (blood routine, blood biochemistry, coagulation function, thyroid function (FT3, FT4, TSH), urinalysis, etc.), and auxiliary examinations (anteroposterior chest X-ray, 12-lead ECG, ultrasonography) with all indices normal or abnormal but without clinical significance.
5. Willing to participate in the planned pharmacokinetic (PK) blood sampling studies and able to comply with the medication and blood sample collection procedures.
6. Negative blood pregnancy test within 24 hours before the first dose, and the participant must agree to use effective contraceptive measures during the study period and for 6 months after medication, agreeing to use at least one of the following contraceptive methods:

Condoms; Subcutaneous contraceptive implant; Intrauterine device or intrauterine system; High-efficiency oral contraceptives, combined or progestin-only; Injectable progestin; Contraceptive vaginal ring; Transdermal contraceptive patch.

Exclusion Criteria:

1. Significant prolongation of QT/QTc interval during the screening period and baseline (e.g., repeatedly confirmed QTcF interval > 450 ms);
2. Organic lesions in vital organs such as the heart, liver, kidneys, brain, and lungs; a clear history of diseases or other significant conditions in the central nervous system, cardiovascular system, cerebrovascular, hematologic, urinary, digestive, respiratory, metabolic, and musculoskeletal systems; a history of autoimmune diseases; a history of endocrine disorders, such as thyroid dysfunction;
3. Diseases of the gastrointestinal tract, liver, kidneys, or other conditions known to interfere with drug absorption, distribution, metabolism, or excretion;
4. Suffering from malignant tumors or any history of any malignancy within 5 years prior to screening (except for completely resected carcinoma in situ of the cervix, non-metastatic cutaneous squamous cell carcinoma, or basal cell carcinoma);
5. Other risk factors for torsades de pointes ventricular tachycardia (TdP) in the medical history (such as heart failure, hypokalemia, family history of long QT syndrome);
6. History of organ transplantation or use of immunosuppressants agents within in the past 3 months or planned use, including but not limited to; calcineurin inhibitors such as tacrolimus and cyclosporine; mycophenolate agents such as mycophenolate mofetil and mycophenolate sodium enteric-coated tablets; glucocorticoids medications such as prednisone and methylprednisolone; others such as sirolimus, azathioprine, mizoribine and leflunomide;
7. History of poorly controlled psychiatric illness with medication;
8. Current or history of severe or persistent infection within the past 3 months (requiring hospitalization or opportunistic infection); or evidence of active and uncontrolled viral infections such as HIV, HBV (HBsAg positive), HCV (anti-HCV antibody positive), syphilis, or any bacterial, parasitic, or fungal infection requiring treatment;
9. Allergy to rhG-CSF products (including rhG-CSF and PEG-modified rhG-CSF) and their components, or allergy to recombinant human proteins or polypeptide drugs derived from Escherichia coli;
10. Use of human granulocyte colony-stimulating factor (G-CSF) therapies within the past 3 months prior to screening; planned or current use of drugs with potential drug interactions with G-CSF therapies, such as lithium;
11. Use of any prescription or over-the-counter medications (including traditional Chinese medicine, health supplements, etc.) within 14 days before the first dose of the test drug or during the drug's 5 half-lives (whichever is longer), unless both the investigator and the sponsor agree that it has no impact on the clinical study;
12. Current or planned use of aspirin, statins, and/or any other drugs that affecting the pathogenesis of preeclampsia (including but not limited to low molecular weight heparin, broccoli sprout extract tablets, digoxin immune Fab, recombinant antithrombin III, proton pump inhibitors, metformin, etc.);
13. Concomitant use with drugs that prolong the QT/QTc interval;
14. Vaccination with live or attenuated vaccines within 3 months before the start of the trial;
15. History of drug abuse, drug use, or alcoholism (drug abuse history or use of narcotics in the past five years; consumption of 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
16. Smoking (or use of tobacco-containing products) in the past 3 months, or unwillingness to refrain from smoking during the study period;
17. Participation in a clinical drug trial within the past 3 months or during the time frame equivalent to 5 times the drug's half-life as specified in other trial drug package inserts/investigator brochures/informed consent forms (whichever is longer), or other conditions deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Adverse Event（AE） | Day1-21.
blood pressure | Day1-21.
pulse | Day1-21.
respiration | Day1-21.
Temperature | Day1-21.
Number of participants with clinically significant change from baseline in physical examination. | Day1-21.
Number of participants with clinically significant change from baseline in laboratory test. | Day1-21.
Number of participants with clinically significant change from baseline in ultrasound imaging. | Day1-21.
Electrocardiogram (including QT/QTc interval) | Day1-21
Anti-drug antibody. | Day1-21
Area under the plasma drug concentration-time curve, AUC 0-t. | Day15,336 hours after dosing.
Area under the plasma drug concentration-time curve from time 0 to infinity, AUC 0-∞. | Day15，336 hours after dosing.
Maximum concentration (Cmax) | Day15，336 hours after dosing.
Time to maximum concentration(Tmax) | Day15，336 hours after dosing.
Drug half-life (t1/2) | Day15，336 hours after dosing.
Clearance (CL/F) | Day15，336 hours after dosing.
Apparent Volume of Distribution (Vd/F) | Day15，336 hours after dosing.

SECONDARY OUTCOMES:
CD34+ cell level | Day21，21 days after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No